CLINICAL TRIAL: NCT01162473
Title: A Study of the Efficacy of Milk Oral Immunotherapy in Children
Brief Title: Milk Oral Immunotherapy in Children to Treat Food Allergy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-007320
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Milk Hypersensitivity
Keywords: Food hypersensitivity; Milk hypersensitivity; Milk allergy; Food allergy
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Sensitivity (Active Comparator): All subjects will undergo a food challenge (week 2). Subjects undergoing delayed desensitization via milk oral immunotherapy with milk protein powder will begin build-up of desensitization during Week 16 and continue thru Week 50. Total active participation will last 51 weeks.
  Interventions: Dietary Supplement: Milk Oral Immunotherapy; Drug: Milk Protein Powder; Other: Food Challenge
- Immediate Sensitivity (Active Comparator): All subjects will undergo a food challenge (week 2). Subjects undergoing immediate desensitization via milk oral immunotherapy with milk protein powder will begin build-up of desensitization during Week 3 and continue thru Week 35. Total active participation will last 38 weeks.
  Interventions: Dietary Supplement: Milk Oral Immunotherapy; Drug: Milk Protein Powder; Other: Food Challenge

INTERVENTIONS:
Dietary Supplement: Milk Oral Immunotherapy — Subjects will participate in a desensitization protocol over the course of 13 weeks to reach a goal maintenance dose of 8 ounces of cow's milk. Once reaching maintenance, subjects will continue on this dose for 12 additional weeks.
Drug: Milk Protein Powder — Milk protein powder will be administered in incremental doses during the desensitization protocol.
Other: Food Challenge

SUMMARY:
Background and Rationale

For patients with Immunoglobulin E (IgE)-mediated food allergy, the current management includes identification of the causative food and avoidance. Specifically, among young children, cow's milk allergy is the most common food allergy, occurring in as many as 2-3%. Given the prevalence of milk and the difficulty to avoid it in the diet, the investigators aim to investigate the safety and efficacy of oral immunotherapy for cow's milk allergy.

Main Objective

The primary objective is to study the efficacy of milk oral immunotherapy.

Target Population

Children aged six to 17 years with a history of cow's milk allergy will be recruited from The Children's Hospital of Philadelphia Allergy clinical offices for the investigators study.

DETAILED DESCRIPTION:
Primary Study Interventions

Prior to and after the desensitization, we will conduct double-blind placebo controlled food challenges to cow's milk protein. During the desensitization phase, we will give increasing doses of cow's milk protein by mouth on a weekly basis, as tolerated. The desensitization protocol starts with dilutional doses of milk and build up to a goal of 8 ounces of cow's milk.

Main Study Outcome Measure

The percentage of children completing the desensitization protocol in each study group will be the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be age six to 17 years and have a history of cow's milk allergy. Subjects shall maintain strict avoidance of consumption of all cow's milk protein containing foods.
2. Subjects will have a history (within the past six months) of a positive skin prick test to milk extract or an immunocap IgE level greater than 0.35 kilounits per liter (kU/L), and a positive allergic reaction history to milk within the past 12 months.
3. Subjects must be in good health, as determined by medical history and physical examination performed by a study physician.
4. Females of childbearing potential must be using an effective method of contraception, including abstinence, and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.
5. Informed consent of parent or legal guardian is required.

Exclusion Criteria:

1. Ability to tolerate eight ounces of cow's milk or eight grams of milk protein powder
2. Pregnancy
3. A history of soy allergy
4. A history of food protein induced enterocolitis syndrome to milk
5. A history of anaphylaxis requiring hospitalization
6. A history of intubation related to asthma and/or a history of an intensive care unit admission for asthma management
7. A current diagnosis of severe persistent asthma [forced expiratory volume in 1 second (FEV1) < 60% of predicted, as defined by National Heart, Lung, and Blood Institute (NHLBI) guidelines, despite current therapy
8. A current diagnosis of severe atopic dermatitis
9. A serious chronic medical condition, including neurologic, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease
10. Use of oral or injection steroids within one month of protocol initial visit
11. An acute illness within one week prior to the first dose of oral immunotherapy
12. Use of antihistamines within seven days prior to double blind placebo controlled food challenge (DBPCFC)
13. Use of chronic immunomodulatory therapy
14. Participation in another experimental therapy study
15. Participation in a study for the treatment of food allergy in the past 12 months
16. Inability to discontinue antihistamines for skin testing and food challenges

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M. Spergel, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia; Antonella Cianferoni, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bollinger ME, Dahlquist LM, Mudd K, Sonntag C, Dillinger L, McKenna K. The impact of food allergy on the daily activities of children and their families. Ann Allergy Asthma Immunol. 2006 Mar;96(3):415-21. doi: 10.1016/S1081-1206(10)60908-8. PMID 16597075
- [Background] Skripak JM, Nash SD, Rowley H, Brereton NH, Oh S, Hamilton RG, Matsui EC, Burks AW, Wood RA. A randomized, double-blind, placebo-controlled study of milk oral immunotherapy for cow's milk allergy. J Allergy Clin Immunol. 2008 Dec;122(6):1154-60. doi: 10.1016/j.jaci.2008.09.030. Epub 2008 Oct 25. PMID 18951617
- [Background] Longo G, Barbi E, Berti I, Meneghetti R, Pittalis A, Ronfani L, Ventura A. Specific oral tolerance induction in children with very severe cow's milk-induced reactions. J Allergy Clin Immunol. 2008 Feb;121(2):343-7. doi: 10.1016/j.jaci.2007.10.029. Epub 2007 Dec 26. PMID 18158176
- [Background] Meglio P, Bartone E, Plantamura M, Arabito E, Giampietro PG. A protocol for oral desensitization in children with IgE-mediated cow's milk allergy. Allergy. 2004 Sep;59(9):980-7. doi: 10.1111/j.1398-9995.2004.00542.x. PMID 15291907
- [Background] Zapatero L, Alonso E, Fuentes V, Martinez MI. Oral desensitization in children with cow's milk allergy. J Investig Allergol Clin Immunol. 2008;18(5):389-96. PMID 18973104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with a history of cow's milk allergy were referred from CHOP Allergy Clinics located in the main campus and satellite offices. Allergy and general pediatric practices in the greater Philadelphia area were also contacted by study staff as part of enrollment outreach.
Groups:
- Delayed Sensitivity: All subjects underwent a food challenge (week 2). Subjects undergoing delayed desensitization via milk oral immunotherapy with milk protein powder began build-up of desensitization during Week 16 and continued thru Week 50. Total active participation lasted 51 weeks.
- Immediate Sensitivity: All subjects underwent a food challenge (week 2). Subjects undergoing immediate desensitization via milk oral immunotherapy with milk protein powder began build-up of desensitization during Week 3 and continued thru Week 35. Total active participation lasted 38 weeks.
Period: Overall Study
Arm/Group | Delayed Sensitivity | Immediate Sensitivity
Started | 8 | 17
Completed | 6 | 12
Not Completed | 2 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Sensitivity | Immediate Sensitivity | Total
Number analyzed (Participants) | 8 | 17 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 17 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.25 [6 to 12] | 8.88 [6 to 13] | 8.68 [6 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 5 | 11 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 17 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Completed Desensitization Protocol
Description: Subjects who withdrew prior to completing the desensitization protocol and those who experienced anaphylaxis during the desensitization protocol (i.e., were unable to complete the protocol) were considered to be "treatment failures". Subjects who completed the desensitization protocol were considered to be "treatment successes".
Time Frame: 1 year
Population: The analysis population included all subjects who began desensitization per protocol.
Measure: Number; unit: participants
Arm/Group | Delayed Sensitivity | Immediate Sensitivity
Number analyzed (Participants) | 8 | 17
participants | 6 | 12

ADVERSE EVENTS:
Time Frame: 1 year
Description: Safety was assessed at all follow-up clinic visits. Adverse events encountered during the previous week, as documented on subjects' event journals, were reviewed. Full physical exams performed and vital signs were obtained. During desensitization, families were contacted every other day (first week) and then twice a week (weeks 2-6).
Groups:
- Delayed Desensitization: Subjects undergoing delayed desensitization via milk oral immunotherapy with milk protein powder (42 week protocol).
- Immediate Desensitization: Subjects undergoing immediate desensitization via milk oral immunotherapy with milk protein powder (29 week protocol)
Arm/Group | Delayed Desensitization | Immediate Desensitization
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/17
Other Adverse Events (participants affected / at risk) | 1/8 | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Desensitization (N=8) | Immediate Desensitization (N=17)
Anaphylaxis (Immune system disorders) | 2 (2) | 1 (1) — 3 subjects required epinephrine
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Desensitization (N=8) | Immediate Desensitization (N=17)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
The small sample size constrains the statistical significance of this study. While useful in indicating potential trends, the results of this pilot study should be cautiously interpreted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No